CLINICAL TRIAL: NCT02753816
Title: The Effect of Tranexamic Acid (TXA) on Blood Loss and Transfusion Rates in Burn Wound Surgery - A Randomized, Double-Blinded Placebo-Controlled Trial
Brief Title: TXA Study in Major Burn Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment and goals unable to be reached.
Sponsor: Corewell Health West (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-154
Record Dates: First submitted 2016-04-18; First posted 2016-04-28 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-04

CONDITIONS: Tranexamic Acid; Burn; Major Surgery
Keywords: Tranexamic Acid; Burn; Surgery; Tangential; Excision
MeSH Terms: conditions — Burns | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tranexamic Acid (Experimental): 1 gram of Tranexamic Acid given over 10 minutes into the vein once prior to surgery
  Interventions: Drug: Tranexamic Acid
- Placebo (Placebo Comparator): Placebo given over 10 minutes into the vein once prior to surgery
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic Acid
Drug: Placebo Comparator
  Arms: Placebo

SUMMARY:
Major surgery can result in blood loss that can require a blood transfusion during and/or after surgery. Tranexamic acid (TXA) is a medication that was first introduced in the 1960's as a treatment for heavy menstrual bleeding. Over the past 20 years, it has been used and studied in patients undergoing open-heart surgery, liver transplantation, and urologic surgery. Investigators believe tranexamic acid may possibly decrease bleeding related to major burn surgery, resulting in reduced blood loss, lower blood transfusion rates, and possibly decreased hospital costs related to your stay.

In this study, prior to each surgical procedure to treat the participants burn injury, the participant will receive either the drug tranexamic acid or placebo. The placebo is a liquid that looks like the tranexamic acid medicine, but does not have any active ingredient in it. In this study, both the tranexamic acid and the placebo are considered research.

DETAILED DESCRIPTION:
Neither the participant nor the study doctor will choose what treatment the participant gets. The participant will have an equal chance of being given the tranexamic acid or the placebo. Neither the participant nor the study doctor will know which treatment the participant is receiving.

The participant will receive one 1 gram dose of either tranexamic acid or placebo immediately before surgery. The dose of tranexamic acid or placebo will be given in the participants vein over a 10-minute period.

Information from the participants medical record related to their surgery and recovery time in the hospital will be collected by medical staff assisting with this study and recorded on study forms. These study forms will be labeled with the participants study number instead of their name.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing burn excision surgery for standard of care purposes (to include: greater than or equal to 350 cm2 of full thickness or deep partial thickness burns)
* Male or female > 18 years of age
* Subject or subject's medical decision maker agrees to participate in this study and provides informed consent

Exclusion Criteria:

* Subjects with a history of hypercoagulopathy, deep vein thrombosis (DVT), pulmonary embolism
* Baseline creatinine level greater than 2.83 mg/dL
* Subjects with known hypersensitivity to tranexamic acid
* Patients with acquired defective color vision
* Patients with subarachnoid hemorrhage
* Children
* Pregnant women
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-04; Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Steensma, MD, Principal Investigator — Corewell Health West
Locations (1):
- Spectrum Health Hospital, Grand Rapids, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Engrav LH, Heimbach DM, Reus JL, Harnar TJ, Marvin JA. Early excision and grafting vs. nonoperative treatment of burns of indeterminant depth: a randomized prospective study. J Trauma. 1983 Nov;23(11):1001-4. doi: 10.1097/00005373-198311000-00007. PMID 6355500
- [Background] Ong YS, Samuel M, Song C. Meta-analysis of early excision of burns. Burns. 2006 Mar;32(2):145-50. doi: 10.1016/j.burns.2005.09.005. Epub 2006 Jan 18. PMID 16414197
- [Background] Desai MH, Herndon DN, Broemeling L, Barrow RE, Nichols RJ Jr, Rutan RL. Early burn wound excision significantly reduces blood loss. Ann Surg. 1990 Jun;211(6):753-9; discussion 759-62. doi: 10.1097/00000658-199006000-00015. PMID 2357138
- [Background] Curinga G, Jain A, Feldman M, Prosciak M, Phillips B, Milner S. Red blood cell transfusion following burn. Burns. 2011 Aug;37(5):742-52. doi: 10.1016/j.burns.2011.01.016. Epub 2011 Mar 1. PMID 21367529
- [Background] Muller M, Gahankari D, Herndon DN. Operative wound management. Total burn care. 2007;3:177-195.
- [Background] Vermylen J, Verhaegen-Declercq ML, Fierens F, Verstraete M. A double blind study of the effect of tranexamic acid in essential menorrhagia. Bull Soc R Belge Gynecol Obstet. 1968;38(5):385-90. No abstract available. PMID 4890296
- [Background] Prentice CR. Basis of antifibrinolytic therapy. J Clin Pathol Suppl (R Coll Pathol). 1980;14:35-40. No abstract available. PMID 6159375
- [Background] Wei W, Wei B. Comparison of topical and intravenous tranexamic acid on blood loss and transfusion rates in total hip arthroplasty. J Arthroplasty. 2014 Nov;29(11):2113-6. doi: 10.1016/j.arth.2014.07.019. Epub 2014 Jul 30. PMID 25155138
- [Background] Patatanian E, Fugate SE. Hemostatic mouthwashes in anticoagulated patients undergoing dental extraction. Ann Pharmacother. 2006 Dec;40(12):2205-10. doi: 10.1345/aph.1H295. Epub 2006 Nov 7. PMID 17090725
- [Background] Mangano DT, Tudor IC, Dietzel C; Multicenter Study of Perioperative Ischemia Research Group; Ischemia Research and Education Foundation. The risk associated with aprotinin in cardiac surgery. N Engl J Med. 2006 Jan 26;354(4):353-65. doi: 10.1056/NEJMoa051379. PMID 16436767
- [Background] Williams-Johnson JA, McDonald AH, Strachan GG, Williams EW. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2) A randomised, placebo-controlled trial. West Indian Med J. 2010 Dec;59(6):612-24. PMID 21702233
- [Background] Jennes S, Degrave E, Despiegeleer X, Grenez O. Effect of tranexamic acid on blood loss in burn surgery: A preliminary study: 33. Journal of Burn Care & Research. 2003;24:S59.
- [Background] Tang YM, Chapman TW, Brooks P. Use of tranexamic acid to reduce bleeding in burns surgery. J Plast Reconstr Aesthet Surg. 2012 May;65(5):684-6. doi: 10.1016/j.bjps.2011.09.028. Epub 2011 Oct 7. PMID 21983540
- [Background] Poeran J, Rasul R, Suzuki S, Danninger T, Mazumdar M, Opperer M, Boettner F, Memtsoudis SG. Tranexamic acid use and postoperative outcomes in patients undergoing total hip or knee arthroplasty in the United States: retrospective analysis of effectiveness and safety. BMJ. 2014 Aug 12;349:g4829. doi: 10.1136/bmj.g4829. PMID 25116268
- [Background] Satahoo SS, Parikh PP, Naranjo D, Davis JS, Duncan RC, Pizano LR, Namias N, Schulman CI. Are burn patients really at risk for thrombotic events? J Burn Care Res. 2015 Jan-Feb;36(1):100-4. doi: 10.1097/BCR.0000000000000093. PMID 25084492
- [Background] Twisk JWR. Applied Multilevel Analysis: A Practical Guide for Medical Researchers. 2006. Cambridge University Press, London, UK.
- [Background] American Burn Association. Burn incidence fact sheet. http://www.ameriburn.org/resources_factsheet.php. Accessed May 20, 2015.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants can have multiple surgeries during the course of their stay. This is the reason for the discrepancy between the protocol enrollment and the participant flow.
Units Other Than Participants: Number of surgeries
Groups:
- Tranexamic Acid: 1 gram of Tranexamic Acid given over 10 minutes into the vein once prior to surgery
  Tranexamic Acid
- Placebo: Placebo given over 10 minutes into the vein once prior to surgery
  Placebo Comparator
- Tranexamic Acid and Placebo: Patients whom received Tranexamic Acid during one surgery and Placebo in another surgery
Period: Overall Study
Arm/Group | Tranexamic Acid | Placebo | Tranexamic Acid and Placebo
Started | 7; 9 Number of surgeries | 11; 11 Number of surgeries | 7; 22 Number of surgeries
Tranexamic Acid | 7; 9 Number of surgeries | 0; 0 Number of surgeries | 7; 12 Number of surgeries
Placebo | 0; 0 Number of surgeries | 11; 11 Number of surgeries | 7; 10 Number of surgeries
Completed | 7; 9 Number of surgeries | 10; 10 Number of surgeries | 7; 22 Number of surgeries
Not Completed | 0; 0 Number of surgeries | 1; 1 Number of surgeries | 0; 0 Number of surgeries
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tranexamic Acid and Placebo: (see participant flow)
- Total: Total of all reporting groups
Arm/Group | Tranexamic Acid | Placebo | Tranexamic Acid and Placebo | Total
Number analyzed (Participants) | 7 | 11 | 7 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 8 | 6 | 21
  >=65 years | 0 | 3 | 1 | 4
Age, Continuous [Mean (Full Range); unit: years] | 37.2 [23.9 to 51.0] | 53.7 [36.1 to 69.9] | 48.6 [33.8 to 74.6] | 47.6 [23.9 to 74.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 1 | 7
  Male | 6 | 6 | 6 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 11 | 7 | 25

OUTCOME MEASURES:

1. Primary Outcome: Intraoperative Blood Loss in mL
Description: To determine the impact of perioperative administration of Tranexamic Acid on blood loss in major burn surgeries.
Time Frame: Intraoperative, average 122 minutes
Population: 1 patient in the Placebo group was excluded from this analysis. Patient was randomized to treatment but never received the treatment intraoperatively. 1 additional patient from the Placebo group was also excluded due to the missing data required to calculate intraoperative blood loss.
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 14 | 15
mL | 100 [100 to 200] | 325 [200 to 500]

2. Primary Outcome: Blood Transfusion Rates, Defined Nominally (Binary) as Having at Least One Transfusion
Description: To determine the impact of perioperative administration of Tranexamic Acid on transfusion rates in major burn surgeries.
Time Frame: First burn surgery to hospital discharge
Population: 1 patient in the Placebo group was excluded from this analysis. Patient was randomized to treatment but never received the treatment intraoperatively. 1 additional patient from the Placebo group was also excluded due the missing data required to calculate transfusion rate . 1 patient from the Tranexamic Acid group was excluded due to missing data required to calculate transfusion rate.
Measure: Number; unit: Patients with 1 or more transfusions
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 13 | 15
Patients with 1 or more transfusions | 2 | 3

3. Secondary Outcome: Effect of Tranexamic Acid on the Total Length of Hospital Admission for a Large (350 cm2) Burn Injury
Description: To determine the impact of Tranexamic Acid on total hospital length of stay by comparing the hospital admission date and the hospital discharge date. This determination will take into account current burn size and location, procedures performed and their effect on wound healing and skin graft survival.
Time Frame: Hospital admission to hospital discharge
Population: For this analysis we compared patients that only received either Tranexamic Acid or Placebo. 3 patients from the Tranexamic Acid group and 2 from the Placebo group were not included in the analysis due to missing data on their length of stay.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Tranexamic Acid | Placebo
Number analyzed (Participants) | 5 | 8
Days | 23 [10 to 29] | 9 [5 to 23]

ADVERSE EVENTS:
Time Frame: Hospital admission to hospital discharge
Arm/Group | Tranexamic Acid | Placebo
All-Cause Mortality (participants affected / at risk) | 1/14 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/14 | 1/17
Other Adverse Events (participants affected / at risk) | 0/14 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tranexamic Acid (N=14) | Placebo (N=17)
NSTEMI (Cardiac disorders) | 0 (0) | 1 (1) — suffered MI (Myocardial Infarction) one day following treatment - MI was determined to be "Severe, Not at all related"
Pulmonary Embolism (Vascular disorders) | 1 (1) | 0 (0) — Suffered PE (Pulmonary Embolism) 3 days following treatment * PE was determined to be "Severe, Unlikely Related"
Acute Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) — Patient suffered an Acute Myocardial Infarction one day after study procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-10): https://cdn.clinicaltrials.gov/large-docs/16/NCT02753816/Prot_SAP_000.pdf